CLINICAL TRIAL: NCT03367728
Title: Randomized, Double-Blinded, Placebo-Controlled Trial to Investigate the Role of Laparoscopic Transversus Abdominis Plane Block in Gastric Bypass Surgery (LapTAP Trial)
Brief Title: The Use of Laparoscopic Transversus Abdominis Plane Block in Gastric Bypass Surgery (LapTAP)
Acronym: LapTAP
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20170749-01H
Record Dates: First submitted 2017-12-05; First posted 2017-12-11 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Bariatric Surgery Candidate
Keywords: Bariatric Surgery; Bariatrics; Ropivacaine; Randomized Controlled Trial; Enhanced Recovery After Bariatric Surgery; TAP Block; Rectus Sheath Block
MeSH Terms: interventions — Ropivacaine; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TAP and Rectus Sheath Normal Saline (Placebo Comparator): TAP and Rectus Sheath Block of 60 mL Normal Saline divided into 4 injections administered as in Experimental Arm.
  Interventions: Drug: Normal saline
- TAP and Rectus Sheath ropivacaine (Experimental): The block will be administered in the anterior abdominal wall. For the TAP block, the standard technique will be followed- at the anterior axillary line midway between the subcostal margin and iliac crest. For the rectus sheath block, a bilateral sub-xiphoid approach will be used. There will be 4 injection sites in total and the size of the needle will be standardized to an 18g spinal needle 10cms. Using laparoscopic visualization, the transversus abdominis muscles were identified lateral to the semilunar line. Ropivacaine to be infiltrated will be divided into 4 equal amounts. The procedure is then repeated 2 times in the transversus abdominis plane (20mL each) and 2 times as a Rectus Sheath Block (10mL each) with a total amount of 60 mL.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — TAP and Rectus Sheath Block Injections of Ropivacaine
  Other Names: NAROPIN®; 84057-95-4
  Arms: TAP and Rectus Sheath ropivacaine
Drug: Normal saline — TAP and Rectus Sheath Block Injections of Normal Saline
  Other Names: Sodium Chloride; 7647-14-5
  Arms: TAP and Rectus Sheath Normal Saline

SUMMARY:
Randomized, Double-Blinded, Placebo-Controlled Trial of Laparoscopic Transverse Abdominis Plane (Lap TAP) and Rectus Sheath Block in elective Gastric Bypass Surgery aiming to evaluate the benefit of a laparoscopically -guided, surgical transversus abdominis plane (TAP) block and rectus sheath block in reducing post-operative opioid consumption and improving outcomes in patients undergoing laparoscopic gastric bypass surgery. The results of this study will provide further evidence on the optimal means to obtain analgesia in patients undergoing gastric bypass surgery

DETAILED DESCRIPTION:
Management of post-operative pain remains a major challenge and an area of continued research. Effective pain control, apart from providing general patient comfort, is critical for a variety of clinical reasons. It leads to early ambulation and improved respiratory function, which significantly reduces the risk of post-operative complications such as pulmonary embolus or pneumonia, as well as early discharge.

Post-operative pain management was typically opioid-based; however, post-operative opioid use may be associated with increased risk of respiratory depression and sedation. It is therefore desirable to implement opioid sparing multimodal analgesia to achieve satisfactory pain control while reducing post-operative opioid requirements and their side-effects.

Rational pain management is a particularly pertinent issue in the patients with morbid obesity (MO). The pathophysiology of obesity, the high prevalence of obstructive sleep apnea, and high susceptibility to respiratory depression amongst patients with MO make safe analgesic (pain) management especially difficult. These individuals are at high risk of post-operative adverse respiratory events, nosocomial infections, cardiovascular complications, and pulmonary emboli (the second leading cause of death in the bariatric surgery population).

Given the increasing number of patients with MO presenting for elective weight loss surgery, it is important to understand and optimize the analgesic requirements of this patient population. However, there are limited evidence-based recommendations and no ideal analgesic regimen exists for patients with MO. Current recommendations include use of step-wise severity-based opioid- sparing multimodal analgesia. It is possible that including local anesthetic blocks will further reduce pain, opioid analgesic consumption and side-effects from pain management (sedation, confusion, nausea & vomiting etc.) at-risk patient population.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing Roux-en-Y gastric bypass surgery;
* Patients who able to tolerate general anesthetic and pneumoperitoneum;
* Patients who able to provide informed consent for the surgery;
* Patients over the age of 18 years;

Exclusion Criteria:

* Patient undergoing planned sleeve gastrectomy (intra-op conversion to sleeve gastrectomy after delivery of Ropivacaine/placebo will be included and analyzed using intention-to-treat approach)
* Patients with an allergy to local anesthetics
* Patients with severe underlying cardiovascular disease (ie: congestive heart failure, conduction abnormalities, and ischemic heart disease)
* Patients with chronic renal disease Stage 3 or greater (Creatinine clearance less than 60mL/min)
* Patients with hepatic dysfunction Child-Pugh Class B or C
* Patients with previous foregut surgery including esophageal, gastric, liver, and pancreas resections
* Patients weighing less than or equal to 100 kilograms as measured in the pre-admission unit
* Patients enrolled in any other study involving involve tissue biopsy.
* Patients with Chronic Pain and Chronic Opioid use- Oral Morphine Equivalent of >100mg/day

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-11-27 (Actual); Primary Completion 2020-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Cumulative postoperative narcotic use | Hour 0-24 post operatively
  Cumulative postoperative narcotic use administered within a max of 24 post operatively

SECONDARY OUTCOMES:
Peak Expiratory flow score | Hour 0-24 post operatively
  measured by the spirometry 60 - 850 liters per minute. Peak expiratory force has not been studied extensively in obese patients. Currently, there is no recommendation on what constitutes a clinically significant change. Recovery to baseline will be sought.
Post-operative pain score | Hour 0-24 post operatively
  measured by the 0-10 Numeric pain rating score
6-minute walk distance (6MWD) | 0-24 Hour post operatively
  the distance (m) an individual is able to walk along a flat 30 m walkway over a six-minute period, with breaks as required
Quality of Life Questionnaire (QOR-40) | 0-24 Hour post operatively
  Assessment of different aspects of quality of life using validated questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Mamazza, MD, Principal Investigator — The Ottawa Hospital
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Within 6 months of completion

REFERENCES:
- [Derived] Jarrar A, Budiansky A, Eipe N, Walsh C, Kolozsvari N, Neville A, Mamazza J. Randomised, double-blinded, placebo-controlled trial to investigate the role of laparoscopic transversus abdominis plane block in gastric bypass surgery: a study protocol. BMJ Open. 2020 Jun 28;10(6):e025818. doi: 10.1136/bmjopen-2018-025818. PMID 32595142